CLINICAL TRIAL: NCT05750784
Title: Personalized Approach to Robotic Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 199731
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; robotic total knee arthroplasty; the active robotic surgical system; kinematic alignment; mechanical alignment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total knee arthroplasty using the active robotic system using the kinematic alignment concept (Other): Total knee arthroplasty using the active robotic surgical system TSolution One TCAT, and system for planning TPlan
  Interventions: Procedure: Total knee arthroplasty using the active robotic surgical system
- total knee arthroplasty using the active robotic system using the mechanical alignment concept (Other): Total knee arthroplasty using the active robotic surgical system TSolution One TCAT, and system for planning TPlan
  Interventions: Procedure: Total knee arthroplasty using the active robotic surgical system

INTERVENTIONS:
Procedure: Total knee arthroplasty using the active robotic surgical system — Total knee arthroplasty using the active robotic surgical system TSolution One TCAT, and system for planning TPlan

SUMMARY:
For the first time in Russia, it is planned to introduce a system of personalized preoperative planning, applying the concept of kinematic alignment in robotic knee arthroplasty. Aim: to improve the results of robotic knee alignment by developing and implementing a personalized approach in preoperative planning. Objectives: to develop a system of personalized robotic knee arthroplasty; implementation of the system in clinical practice, to determine indications, contraindications; study of the results of personalized endoprosthetics, comparison with the results of mechanical alignment; detection of complications; development of an algorithm and protocol for personalized endoprosthetics. It is planned to conduct an open retrospective and prospective clinical study in parallel groups. The study is planned to include 150 patients with osteoarthritis of the knee joint stage 3-4 (according to Kellgren-Lawrence). The methodology developed and improved in the dissertation will be introduced into the work of the clinical Departments of Traumatology, Orthopedics and Disaster Surgery, studying the learning curve.

DETAILED DESCRIPTION:
Relevance: Currently, there are 2 main concepts of total knee arthroplasty: mechanical and kinematic alignment of the axis of the lower limb. Mechanical alignment was first proposed by Install JN. It implied the standardization of equipment and tools, the reconstruction of the mechanically neutral axis of the limb. However, the number of patients dissatisfied with the result of endoprosthetics remained high. Bellemans' work argues that for many patients, a mechanically neutral axis of the lower limb is not the normal. This is how the concept of kinematic alignment appeared, the main idea of which was to create an absolutely balanced joint throughout the entire volume of movements and recreate the true levels of articular lines of the joint, before the onset of osteoarthritis. However, the use of standard tools and manual techniques does not allow the full use of this concept. Robotic surgery has the main advantage over manual techniques in the high accuracy of implant positioning and allows you to calculate the mechanical axis and the level of the articular line with high accuracy at the stage of preoperative preparation. The introduction of personalized programs, implants in knee arthroplasty, together with the use of active robotic technology, can restore the individual anatomy and function of the lower limb, which will improve the results of endoprosthetics and reduce the percentage of patients dissatisfied with the operation.

The novelty of the proposed topic: For the first time in Russia, it is planned to introduce a system of personalized preoperative planning, applying the concept of kinematic alignment in robotic knee arthroplasty.

Aim and objectives of the research:

Aim: To improve the results of robotic knee alignment by developing and implementing a personalized approach in preoperative planning.

Objectives: to develop a system of personalized robotic knee arthroplasty; implementation of the system in clinical practice, to determine indications, contraindications; study of the results of personalized endoprosthetics, comparison with the results of mechanical alignment; detection of complications; development of an algorithm and protocol for personalized endoprosthetics.

Type of new research: an open-label, retrospective and prospective observational clinical study in parallel groups.

Research object and number of observations: the study is planned to include 150 patients with osteoarthritis of the knee joint of stage 3-4 (according to Kellgren-Lawrence).

Methods of the research:

1. General clinical examination of patients (collection of complaints, examination, assessment of physical findings and local status);
2. Assessment of the range of motion in the knee joint before and after surgery;
3. Performing X-ray images and CT of the knee joint before and after surgery, with the determination of the angles: HKA, LDFA, MPTA, Q; Preoperative 3D planning on the TPLAN workstation; Surgical treatment. 1) Primary total knee arthroplasty using the active robotic surgical system TSolution One, TCAT, using the concept of kinematic alignment; 2) Primary total knee arthroplasty using the active robotic surgical system TSolution One, TCAT, using the concept of mechanical alignment.

Evaluation of patient treatment results according to scales: VAS, KSS, OKS, WOMAC, ASA, FJS-12.

Methods of statistical processing of the material: statistical processing of data is planned to be carried out on a personal computer using Excel software packages and using standard methods of variation statistics using SPSS 16 statistical software packages.

Estimated research result:

For the first time in Russia, an active robotic system will be introduced into clinical practice using the concept of personalized endoprosthetics for primary total knee .

Indications for the use of this algorithm in patients with osteoarthritis of the knee joint will be determined.

The methodology of preoperative planning will be improved. The results of the initial personalized total knee replacement with the use of an active robotic system will be evaluated.

The methodology developed and improved in the dissertation will be introduced into the work of the clinical bases of the Department of Traumatology, Orthopedics and Disaster Surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of written informed consent of the patient to participate in the study;
2. Patients with stage 3-4 osteoarthritis of the knee joint (according to Kellgren-Lawrence).
3. Men and women from 21 to 90 years old.
4. Pain in the knee joint above 3 points according to VAS
5. Opportunity for observations during the entire study period (12 months);
6. Mental adequacy, ability, willingness to cooperate and to fulfill the doctor's recommendations.

Exclusion Criteria:

1. Refusal of the patient from surgical treatment;
2. Presence of contraindications to surgical treatment;
3. Severe forms of diabetes mellitus (glycosylated hemoglobin> 9%);
4. Diseases of the blood (thrombopenia, thrombocytopenia, anemia with Hb <90 g / l);
5. The patient's unwillingness to conscious cooperation.
6. Refusal of the patient to participate in the study;
7. Non-compliance with the hospital regimen, according to the order of the Ministry of Health and Social Development of Russia dated 01.08.07, No. 514;
8. The impossibility of observing the patient within the control period after the operation.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Implant position assessment | 2 months after surgery
  CT scanning; these diagnostic methods assess the position of the implant, analysis of deformation, assessment of the angles in the knee joint (LDFA, MPTA, MA, these diagnostic methods assess the position of the implant, analysis of deformation, assessment of the angles in the knee joint, analyze the rotation of implant)
Implant position assessment | 6 months after surgery
  CT scanning
Implant position assessment | 12 months after surgery
  CT scanning

SECONDARY OUTCOMES:
Quality of life and knee function assessment | 2,6,12 months after surgery
  Knee Society Score(KSS score), which combines subjective and objective information and separates the knee score (pain, stability, range of motion etc.) from the functional score of the patient (ability to walk, go up and down stairs)
Quality of life assessment (joint awareness after surgery) | 2,6,12 months after surgery
  FJS-12, measures the clinical outcomes focusing on joint awareness after surgery
Quality of life assessment (the condition of patients) | 2,6,12 months after surgery
  WOMAC score is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints
Pain assessment | 2,6,12 months after surgery
  Visual Analog Score (VAS) for pain - dynamics pain assessment
Quality of life assessment (an individual's activities of daily living) | 2,6,12 months after surgery
  OKS score. The OKS is a patient reported outcome measure that consists of 12 questions about an individual's activities of daily living and how they have been affected by pain over the preceding four weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University clinical hospital №1 I.M.Sechenov First Moscow State Medical University. The Department of Traumatology, Orthopedics and Disaster Surgery, Moscow, Russia

REFERENCES:
- [Background] LYCHAGIN A.V.1, a, GRITSYUK A.A.1, b, RUKIN Y.A.1, c, ELIZAROV M.P.1, d, THE HISTORY OF THE DEVELOPMENT OF ROBOTICS IN SURGERY AND ORTHOPEDICS (LITERATURE REVIEW). 2020; 1 (39)2020: 10.17238/issn2226-2016.2020.1.13-19
- [Background] LYCHAGIN A.V. 1, a, RUKIN Y.A. 1, b, GRITSYUK A.A. 1, c, ELIZAROV M.P. 1, d, FIRST EXPERIENCE OF USING AN ACTIVE ROBOTIC SURGICAL SYSTEM IN TOTAL KNEE ARTHROPLASTY. 2019; 4 (38) 2019: 10.17238/issn2226-2016.2019.4.27-33